CLINICAL TRIAL: NCT05510492
Title: The Effect of Training on Intramuscular Injection Practice Given to Nurses on Determining the VG Site, Using the Air Lock and Z Technique: A Randomized Controlled Trial
Brief Title: Effect of Training on IM Injection Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nazike Duruk (Other)
Responsible Party: Sponsor-Investigator, Nazike Duruk, Associate Professor Doctor, PhD, Eskisehir Osmangazi University
Organization: Eskisehir Osmangazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EskisehirAG
Record Dates: First submitted 2022-08-08; First posted 2022-08-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Injections
Keywords: ventrogluteal; intramuscular; injection; nursing
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Evaluation of the skill training given to nurses on intramuscular injection with the z technique from the ventrogluteal region
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): EXPERIMENTAL GROUP CONSISTS OF 47 NURSES.
  Interventions: Other: EDUCATION; Other: APPLIED EDUCATION
- CONTROL GROUP (Experimental): CONTROL GROUP CONSISTS OF 48 NURSES.
  Interventions: Other: EDUCATION

INTERVENTIONS:
Other: EDUCATION — THE EXPERIMENT GROUP WAS GIVEN THEORETICAL AND APPLIED EDUCATION,
  Other Names: THEORETICAL EDUCATION, PRACTICAL TRAINING
Other: APPLIED EDUCATION — the injection was applied on the model by the researcher with the demonstration method according to the "Procedure Steps of Intramuscular Injection with the Z Technique from the Ventrogluteal Region". This process was first ensured by the nurses, and then
  Other Names: demonstration method
  Arms: EXPERIMENTAL GROUP

SUMMARY:
The aim of this study is to observe how many nurses perform the steps of creating an air lock, identifying the ventrogluteal site, and applying the Z-track technique in intramuscular injections after theoretical and practical training.

Research Hypotheses

* The rate of administering intramuscular injections into the ventrogluteal site will be higher in the intervention group that receives low-fidelity simulator-based training compared to the control group.
* The rate of applying the air-lock technique will be higher in the intervention group that receives low-fidelity simulator-based intramuscular injection training compared to the control group.
* The rate of applying the Z-track technique will be higher in the intervention group that receives low-fidelity simulator-based intramuscular injection training compared to the control group.

DETAILED DESCRIPTION:
This research was designed as a randomized controlled experimental study to observe the extent to which nurses perform the steps of creating an air lock, identifying the ventrogluteal site, and applying the Z-track technique in intramuscular injections after receiving theoretical and practical training.

ELIGIBILITY:
Inclusion criteria:

• Nurses working in inpatient services other than emergency, outpatient clinic, operating room and pediatrics of a Health Practice and Research Hospital

Exclusion Criteria:

• Nurses who do not agree to participate in the research and/or want to leave the research while it is continuing

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
In the study, the effectiveness of the skill training given to nurses was measured. | Since the research was in the pre-test post-test design and the post-test was applied at least two weeks later, the data were collected in a period of up to four months.
  In the evaluation, the observation form of the intramuscular injection procedure steps with the Z technique from the Ventrogluteal region was used. After the trainings, the Student Satisfaction and Self-Confidence in Learning Scale was used. The highest total score that can be obtained from the Student Satisfaction and Self-Confidence in Learning Scale is 65 and the lowest is 13. The high score that can be obtained from the total of the scale indicates high satisfaction and self-confidence. Since the reliability coefficients of the Student Satisfaction and Self-Confidence in Learning Scale and its sub-dimensions vary between 0.826 and 0.914, the scale was found to be reliable.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskişehir Osmangazi Üniversitesi Sağlik, Uygulama Ve Araştirma Hastanesi, Eskişehir, Eski̇şehi̇r, Turkey (Türkiye)

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT05510492/Prot_SAP_000.pdf